CLINICAL TRIAL: NCT00780221
Title: CRP Gene Variants and Coronary Artery Disease in a Chinese Han Population
Brief Title: C-Reactive Protein (CRP) Gene Variants and Coronary Artery Disease in a Chinese Han Population
Acronym: CRP-Han
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Zhongshan Hospital, Shanghai Institute of Cardiovascular Disease,Zhongshan Hospital
Other Study IDs: ZSJQ-30725036; 30725036
Record Dates: First submitted 2008-10-24; First posted 2008-10-27 (Estimated); Last update posted 2008-10-27 (Estimated); Status verified 2008-10

CONDITIONS: Coronary Artery Disease
Keywords: CRP; coronary artery disease; polymorphisms
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sample will be examined and DNA variants be analyzed.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- control: patients without coronary artery disease
- case: patients with coronary artery disease

SUMMARY:
The recognition of the association between circulating C-reactive protein (CRP) levels and risk of coronary heart disease (CHD) has led to an increased emphasis on CRP genetic effects on CRP level and CHD. However, the causality of CRP variants remains uncertain.The objective of this study is to evaluate the association of CRP gene variants and CRP levels in CHD in Chinese Han population. We conduct case-control study in CRP-Han study participants. The common single-nucleotide polymorphisms (SNPs) in the CRP gene, haplotypes, and plasma CRP levels are detected. A Mendelian randomization analysis will be used to help test the likelihood of causal association of gene-CRP levels, CRP levels-CHD and gene-CHD. The investigators hypothesize that CRP gene variants influence the protein level and may participate in CHD progress.

DETAILED DESCRIPTION:
CHD patients and non-CHD population are recruited. CRP level and CHD severity by coronary angiograph will be examined. Mendelian randomization analysis are taken to analyze statically.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of coronary artery disease

Exclusion Criteria:

* with major organ disfunction or acute inflammatory disease

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: in-hospital patients and community healthy individual
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2008-10; Primary Completion 2010-10 (Estimated); Study Completion 2010-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Junbo Ge, Study Director — Shanghai Zhongshan Hospital
Locations (1):
- Zhongshan Hospital, Shanghai, Shanghai Municipality, China